CLINICAL TRIAL: NCT04943185
Title: SLX vs Ab Interno XEN
Brief Title: A Prospective, Single Surgeon, Randomized Control Study Comparing ab Interno XEN Gel Microstent Implantation vs Closed Conjunctiva ab Externo Implantation Performed at the Slit Lamp for the Treatment of Uncontrolled Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de l'oeil des Laurentides (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2018-10526
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: The Objective of the Study is to Prospectively Compare the Success Rate of ab Externo and Interno Implantation

STUDY DESIGN:
Intervention Model Description: The XEN gel stent (Allergan inc.) is a gelatin stent that has been developed for the surgical treatment of medically uncontrolled glaucoma and allows the filtration of aqueous humour from the anterior chamber to the subconjunctival space. The ab interno placement and outcomes of the XEN implant has been described (1,2,3). We describe an ab externo approach to implant the XEN microstent; ab externo closed conjunctiva implantation. This approach has many potential advantages over the ab interno technique, notably a quicker procedure, a potentially better subconjunctival placement of the implant and cost effectiveness due to absent need to rely on an operating room to perform the procedure as it can be done in an office setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ab interno technique (Other): Ab Interno is traditional method of stent XEN implantation, where the device will injected through a small corneal incision that closes with the preloaded XEN injector.
  Interventions: Device: XEN gel microstent implantation
- Ab externo technique (Other): The ab externo approach does this without any incision, less invasive, and the implant is directly injected through the conjunctiva into the anterior chamber of the eye. Both methods create a new way out through the subconjunctival space, which is the traditional target of trabeculectomy.
  Interventions: Device: XEN gel microstent implantation

INTERVENTIONS:
Device: XEN gel microstent implantation — Two differents implantation :
  Ab interno : Operative intervention Ab externo : Slit lamp intervention

SUMMARY:
The objective of the study is to prospectively compare the success rate of ab externo implantation and outcome measures of glaucoma filtering surgery namely IOP (intraocular pressure), number of glaucoma medications, adjunct procedure and adverse events rate compared to the traditional ab interno implantation technique.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE The XEN gel stent (Allergan inc.) is a gelatin stent that has been developed for the surgical treatment of medically uncontrolled glaucoma and allows the filtration of aqueous humour from the anterior chamber to the subconjunctival space. The ab interno placement and outcomes of the XEN implant has been described (1,2,3). We describe an ab externo approach to implant the XEN microstent; ab externo closed conjunctiva implantation. This approach has many potential advantages over the ab interno technique, notably a quicker procedure, a potentially better subconjunctival placement of the implant and cost effectiveness due to absent need to rely on an operating room to perform the procedure as it can be done in an office setting.

Ab interno technique Approximately 6 mm long and as wide as a human hair, this soft gelatinous stent is implanted via an ab interno surgical approach through a small, self-sealing corneal incision, to facilitate aqueous humor drainage from the anterior chamber to the subconjunctival space. The gelatin imparts hydrophilic properties that allow the Gel Implant to conform to the ocular tissue by expanding when hydrated upon contact with the aqueous humor. This expansion might minimize issues such as migration, erosion, and corneal endothelial damage observed in stents with synthetic materials. The ab interno surgical approach for XEN is less invasive than traditional glaucoma surgeries and has several other advantages, including minimal trauma to the conjunctiva, maintenance of the natural drainage pathways, reduced scarring response, and the ability to accurately place the device under direct visualization of anatomy. Minimizing damage to the conjunctiva allows the possibility of future glaucoma surgery. Ab externo technique The transconjunctival ab externo technique is modification of the ab interno procedure. Topical anesthesia with tetracaine 0.5% eye drops is performed before the ocular surface is disinfected with 5% povidone iodine drops. A full blade speculum was used to retract the patient's eyelid, and the patient was positioned at the slit lamp. While the patient gazed down toward the nose, a mixture of an antimetabolite, lidocaine, and epinephrine was injected in the exposed surgical site of the superotemporal quadrant. The antimetabolite is mitomycin C (MMC). The mixture contained either 0.1 cc of MMC (0.2 mg/ml) and 0.05 cc of 2% lidocaine with epinephrine, for a total volume of 0.15 cc. The speculum was then removed. After 5 to 7 minutes, topical anesthesia and disinfection were repeated, and the speculum was secured again. An inserter with a preloaded gel stent is directed to enter the conjunctiva approximately 2 to 3 mm lateral to the intended scleral entry point, and 6 to 7 mm from the limbus, using an aseptic no-touch technique. The inserter was then directed downward to enter the sclera 2.5 mm posterior to the limbus. Once the tip of the inserter needle was visualized in the AC, the plunger of the inserter was advanced while the inserter needle was slowly and simultaneously withdrawn until the gel stent was fully released. The ideal target position of the stent is approximately 3 mm within the subconjunctiva, 2 mm within the sclera, and 1 mm within the AC.

The positioning of the stent was considered successful if a connection was made by the stent between the subconjunctival space and the AC, and a bleb formed. Gonioscopy was performed to confirm proper seating of the gel microstent and slit lamp biomicroscopy was performed to confirm a formed bleb.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with maximally tolerated medically treated (MTMT) uncontrolled glaucoma (POAG, PEX G, PDS G)
2. Male or female who was in good general health and >18 years of age at the time of the preoperative exam
3. The subject complied with post-operative instructions and made their scheduled office appointments

Exclusion Criteria:

Non-Ocular

1. Known or suspected allergy or sensitivity to any medications/diagnostic agents (eg, topical anesthetic, dilating drops, fluorescein) required for this protocol or any of the XEN components (eg, porcine products or glutaraldehyde)
2. Known history of bleeding disorder or prolonged bleeding after surgery (in the opinion of the investigator) or those on pharmacologic blood thinners other than aspirin (up to 100 mg/day)
3. Chemotherapy for cancer treatment within 6 months of screening
4. History of dermatologic keloid formation
5. Participation in another drug/device/observational clinical trial concurrently or concluding within 30 days of screening
6. Any condition that would preclude the patient's ability to comply with study requirements, including completion of the study
7. Any condition or a situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study Ocular
8. Close-angle glaucoma (previous iridotomy laser accepted) active acute angle closure attack, secondary glaucomas (eg, anterior subluxation of the lens, iris or ciliary body cysts, active iris and angle neovascularization, iridocorneal endothelial syndrome,) in the study eye
9. History of following surgeries in the study eye:

   1. incisional refractive surgery (eg, radial keratotomy), other than astigmatic keratotomy or limbal relaxing incisions
   2. corneal graft including partial grafts such as Descemet's stripping endothelial keratoplasty and Descemet's membrane endothelial keratoplasty
   3. previous laser SLT or incisional intraocular surgery that might interfere with the outcome of this trial less than 6 weeks prior to XEN surgery However, previous incisional and laser glaucoma surgeries (eg, trabeculectomy, glaucoma shunt implantation, laser trabeculoplasty, iridotomy, cilioablative procedures) or uncomplicated phacoemulsification with IOL, occurring more than 6 weeks prior to screening, are allowed in the study eye.
10. Previous glaucoma shunt implantation in the target quadrant in the study eye
11. Anticipated need for ocular incisional and/or laser surgery in the study eye during the 12-month follow-up period
12. Ocular (in the study eye) or systemic corticosteroid use within 30 days prior to screening (continuing chronic systemic corticosteroid use is allowed) or known corticosteroid responder
13. Clinically significant inflammation or infection in either eye within 30 days prior to screening (eg, blepharitis, conjunctivitis, keratitis, herpes simplex infection)
14. Active or history of chronic uveitis in the study eye
15. Corneal or other ocular abnormalities (eg, bullous keratopathy, keratoconus) in the study eye that would preclude accurate readings with an applanation tonometer and/or a contact pachymeter, or could confound study results
16. Nanophthalmos in either eye
17. Central corneal thickness ≤ 460 microns or ≥ 620 microns in the study eye
18. Unable to discontinue contact lens wear in the study eye during the studyrevised 2021-03-09 page 6 of 10 protocol: SLX
19. Impaired episcleral venous drainage (eg, Sturge-Weber or other evidence of elevated venous pressure) in the study eye
20. Aphakia, anterior chamber intraocular lens, or previous complicated phacoemulsification surgery in the study eye
21. Vitreous present in the anterior chamber in the study eye
22. Presence of intraocular silicone oil in the study eye
23. Active diabetic retinopathy, choroidal neovascularization, branch retinal vein occlusion, central retinal vein occlusion, proliferative retinopathy, or other ophthalmic disease or disorder in the study eye that could confound study results
24. Female patients who are pregnant, nursing, or planning a pregnancy during the study, or who are of childbearing potential and not using a reliable means of contraception during the study.

For purposes of this study, females will be considered of childbearing potential unless they are naturally postmenopausal or permanently sterilized (ie, tubal occlusion, hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy). Natural menopause is defined as the permanent cessation of menstrual periods, determined retrospectively after a woman has experienced 12 months of amenorrhea without any other obvious pathological or physiological cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Compared the success of interno / externo implantation | 15 minutes by implantation
  The objective of the study is to prospectively compare the success rate of ab externo implantation and outcome measures of glaucoma filtering surgery namely IOP (intraocular pressure), number of glaucoma medications, adjunct procedure and adverse events rate compared to the traditional ab interno implantation technique

CONTACTS AND LOCATIONS:
Locations (1):
- Institutdeloeil, Boisbriand, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
See after the study